CLINICAL TRIAL: NCT06907862
Title: The SWITCH (Substitution of High With Low Ultra-processed Soy Protein Foods In a Guideline-based Diet inTervention for Cardiometabolic Health) Trial
Acronym: SWITCH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Laura Chiavaroli, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB #44955
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Hypertension in Type 2 Diabetes; Diabetes Mellitus Type 2; Dyslipidemia; Hypertension; Metabolic Health; Cardiovascular Risk Factors
Keywords: Randomized controlled trial; Hypertension; Cardiometabolic health; Ultra processed food; technology-based dietary intervention; dehydrated vegetable and fruit blend
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician will be blinded to the nature of the treatment when analyzing data (i.e., will not know the treatment assignment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- enhanced digital dietary intervention (High-UPF soy protein foods) (Active Comparator): The Active Treatment is an enhanced digital dietary intervention with high-UPF soy-containing foods.
  Interventions: Other: Active Treatment
- enhanced digital dietary intervention (Low-UPF soy protein foods) (Active Comparator): The Reference Treatment is an enhanced digital dietary intervention with low-UPF soy-containing foods
  Interventions: Other: Reference Treatment
- Standard of care (Placebo Comparator): usual care provided by their primary care physician and/or specialist
  Interventions: Other: Control

INTERVENTIONS:
Other: Reference Treatment — ≥4 servings/day of soy products categorized as non-ultra processed according to the NOVA classification system (NOVA non-Group 4): ≥2 servings/day of a Group 1 soy milk and ≥1 serving/day of another Group 1 food, such as edamame or roasted soy nuts, and ≥1 serving/day of a Group 3 food, such as tofu or tempeh) as part of a digital dietary intervention, enhanced with 10 servings of vegetables and fruit (5 as dietary advice and 5 provided in a blend of dehydrated vegetables and fruit)
  Arms: enhanced digital dietary intervention (Low-UPF soy protein foods)
Other: Control — Usual care provided by their primary care physician and/or specialist.
  Arms: Standard of care
Other: Active Treatment — ≥4 servings/day of soy products categorized as ultra processed according to the NOVA classification system (NOVA Group 4): ≥2 servings/day of soy milk and ≥2 servings/day of other soy-based products such as soy yogurt, soy burgers, or soy ground round) as part of a digital dietary intervention, enhanced with 10 servings of vegetables and fruit (5 as dietary advice and 5 provided in a blend of dehydrated vegetables and fruit)
  Arms: enhanced digital dietary intervention (High-UPF soy protein foods)

SUMMARY:
This is a randomized, controlled, parallel study with 3 experimental arms aimed to assess the effect of a digital dietary intervention (web-based app, online behavior change curriculum) enhanced with 10 servings of vegetables and fruit (5 as dietary advice within the app, 5 within a dehydrated vegetable and fruit blend), with or without high Ultra Processed Food (UPF) soy-containing proteins compared to standard of care (usual care) on systolic blood pressure (SBP; primary outcome), and other key cardiometabolic endpoints over 12-weeks in adults living with hypertension and obesity, 50% with type 2 diabetes. The main questions this study aims to answer are:

1. Are nutrient-dense, high-UPF soy-protein foods similar (non-inferior) to low-UPF soy-protein foods in the context of a guidelines-based diet in their effect on blood pressure and other cardiometabolic risk factors?
2. Does an enhanced digital dietary intervention lead to meaningful reductions in blood pressure and other cardiometabolic risk factors compared to standard of care?

Participants who are eligible and consent to be part of this study will be randomized to one of the following groups: 1) Active treatment (high-UPF soy-containing enhanced digital dietary intervention), 2) Reference treatment (low-UPF soy-containing enhanced digital dietary intervention), or 3) Control (standard of care).

Participant Requirements:

During the 12-week intervention, all participants will be required to attend in-person clinic visits at baseline (week 0), week 8 and 12.

Baseline Visit (Week 0): Participants will be asked to arrive in a fasted state (no food or beverages, except water, for 10-12 hours before the visit).

* Undergo various assessments, including anthropometric measurements, office blood pressure readings, and blood sampling (via a capillary finger prick and blood sample taken by the study nurse).
* Review the 7-day food records completed using the Keenoa mobile app one week prior to clinic visit.
* Bring fecal and urine samples from home.
* Complete and review all questionnaires received via email one week prior.

Telephone Check-in (Week 1):

One week after beginning the study, the study staff will call participants to check in on how participants are following the protocol and answer any questions.

Mid-Study Visit (Week 8): Participants will be asked to arrive in a fasted state (no food or beverages, except water, for 10-12 hours before the visit).

* Have their office blood pressure and anthropometric measurements taken.
* Complete and review all questionnaires received via email one week prior
* Review the 3-day food records completed using the Keenoa mobile app one week prior to clinic visit.

Final Study Visit (Week 12): Participants will be asked to arrive in a fasted state (no food or beverages, except water, for 10-12 hours before the visit).

* Undergo various assessments, including anthropometric measurements, office blood pressure readings, and blood sampling (via a capillary finger prick and blood sample taken by the study nurse).
* Review the 7-day food records completed using the Keenoa mobile app one week prior to clinic visit.
* Bring fecal and urine samples from home.
* Complete and review all questionnaires received via email one week prior.

Throughout the study, participants will be asked to continue their usual lifestyle and physical activity.

Additional Requirements for Treatment Groups:

Participants randomized to the active and reference treatment groups will also be required to:

* Incorporate a study vegetable and fruit blend (provided) into their daily diet for the full 12 weeks
* Consume soy products categorized as either high ultra processed soy foods at least 4 servings per day, including at least 2 servings of ultra processed soy milk and 2 servings of other soy-based products (e.g., soy yogurt, soy burgers, or soy ground round) or non-ultra processed soy foods at least 4 servings per day, including at least 2 servings of minimally processed soy milk, 1 serving of edamame or roasted soy nuts, and 1 serving of tofu or tempeh
* Participate in the digital dietary intervention, which includes: a health app, 7-day Kickstart Package, weekly text message support, and a 7-session online interactive program designed based on behaviour change theory
* Attend a virtual focus group at Week 4 and complete an online feedback questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Obesity (BMI and waist circumference using sex and ethnic-specific thresholds for obesity and significant abdominal adiposity)
* adults (≥18years)
* hypertension (SBP 130-160 mmHg)
* on stable antihypertensive, antihyperglycemic, antihyperlipidemic, or anti-obesity medications (≥3-months)
* not planning new weight loss for the duration of the trial
* 50% living with type 2 diabetes, HbA1c 6.5-9.0%

Exclusion Criteria:

* Individuals with a history of major cardiovascular events in the last year (stroke or myocardial infarction)
* type 1 diabetes diagnosis
* recent weight loss (≥5 kg over <6 months)
* current treatment with insulin
* eating disorders; substance abuse disorders
* serious depression or psychiatric disorders
* bariatric or recent surgery (<6 months)
* uncontrolled hypertension (SBP/DBP >160/100 mmHg)
* angina pectoris
* gastrointestinal and malabsorption disorders (i.e. inflammatory bowel disease, celiac), pancreatitis, chronic kidney or liver disease, cardiac condition that compromises normal function (e.g. mitral valve disease, heart failure), major disability or disorder requiring continuous medical attention.
* herb or supplement use that may affect primary outcome.
* alcohol use >3 drinks/day; participation in another trial.
* allergies/intolerances to soy; allergies/intolerances to tree nuts, peanuts and seeds (the combination of all 3).
* chronic or prescribed use of medications including prescription NSAIDs, antacids, warfarin, medications affecting NO synthesis (i.e. sildenafil, organic nitrates, etc)
* acute or chronic infection (e.g. active HIV, TB, COVID-19, chronic inflammatory infections such as rheumatoid arthritis)
* use of antibiotics within 3-months of the study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-07 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure | from enrollment to the end of treatment at 12 weeks
  Difference in mean change from baseline.

SECONDARY OUTCOMES:
Key Secondary Outcome: non-high-density lipoprotein cholesterol [non-HDL-C] | from enrollment to the end of treatment at 12 weeks
  Difference in mean change from baseline.
Body weight | from enrollment to the end of treatment at 12 weeks
  Difference in mean change from baseline.
Diastolic Blood Pressure | from enrollment to the end of treatment at 12 weeks
  Difference in mean change from baseline.
Blood Pressure Targets | from enrollment to the end of treatment at 12 weeks
  Difference in proportion achieving therapeutic targets for blood pressure (SBP<140mmHg and DBP <90mmHg for those without diabetes; SBP <130mmHg and DBP <80mmHg for those with diabetes; SBP <120mmHg for Hypertension Canada high-risk patients)
Blood Lipids | from enrollment to the end of treatment at 12 weeks
  Difference in mean change in low-density lipoprotein-cholesterol (LDL-C), triglycerides, and high-density lipoprotein-cholesterol (HDL-C) from baseline.
Blood Lipid Targets | from enrollment to the end of treatment at 12 weeks
  Difference in proportion achieving therapeutic targets for lipids (non-HDL-C <2.6mmol/L, LDL-C <2.0mmol/L)
Glycemic control | from enrollment to the end of treatment at 12 weeks
  Difference in mean change in HbA1c from baseline.
Glycemic control | from enrollment to the end of treatment at 12 weeks
  Difference in mean change in fasting glucose from baseline.
Insulin | from enrollment to the end of treatment at 12 weeks
  Difference in mean change in fasting insulin from baseline.
Insulin Resistance | from enrollment to the end of treatment at 12 weeks
  Difference in mean change in insulin resistance (HOMA-IR) from baseline.
Inflammation | from enrollment to the end of treatment at 12 weeks
  Difference in mean change in C-Reactive Protein (CRP) from baseline.
Body Composition | from enrollment to the end of treatment at 12 weeks
  Difference in mean change in body mass index from baseline.
Body Composition | from enrollment to the end of treatment at 12 weeks
  Difference in mean change in waist circumference from baseline.
Body Composition | from enrollment to the end of treatment at 12 weeks
  Difference in mean change in body fat from baseline.

OTHER OUTCOMES:
Exploratory mechanistic endpoint - DNA Methylation | from enrollment to the end of treatment at 12 weeks
  Difference in mean change from baseline in DNA methylation.
Exploratory mechanistic endpoint - Telomere Length | from enrollment to the end of treatment at 12 weeks
  Difference in mean change from baseline in telomere length.
Exploratory mechanistic endpoint - Intestinal Permeability | from enrollment to the end of treatment at 12 weeks
  Difference in mean change from baseline in intestinal permeability.

CONTACTS AND LOCATIONS:
Locations (1):
- C. David Naylor Building, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All outcomes listed will be shared in an anonymous/de-identified format.
Supporting Information: Study Protocol
Time Frame: IPD and supporting information will be available after the anticipated study completion date from June 2028 and will remain for 30 years until January 2058.
Access Criteria: IPD data will be accessible though the University of Toronto Dataverse (https://borealisdata.ca/dataverse/toronto). The metadata record of our dataset will be public, however access to the data will be restricted. Users will need to request access using the contact information provided in order to view and download our restricted files.